CLINICAL TRIAL: NCT02944864
Title: Phase I Study of Tolerance and Pharmacokinetics of TQ-B3395 in Patients With Advanced Cancer
Brief Title: A Phase I Study of TQ-B3395 on Tolerance and Pharmacokinetics
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Per sponsor request.
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQ-B3395-I-0001
Record Dates: First submitted 2016-10-24; First posted 2016-10-26 (Estimated); Last update posted 2024-09-23 (Actual); Status verified 2016-12

CONDITIONS: Advanced Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQ-B3395 (Experimental): TQ-B3395 QD po and it should be continued until disease progression or intolerable toxicity or patients withdrawal of consent
  Interventions: Drug: TQ-B3395

INTERVENTIONS:
Drug: TQ-B3395 — TQ-B3395 p.o. qd

SUMMARY:
To study the pharmacokinetic characteristics of TQ-B3395 in the human body, recommend a reasonable regimen for subsequent research.

ELIGIBILITY:
Inclusion Criteria:

* Histological documentation of Advanced solid tumors,lack of the standard treatment or treatment failure.In expanding stage,enroll the Non-small Cell Lung Cancer with EGFR+(except exon 20)
* 18-70 years,ECOG PS:0-1,Life expectancy of more than 3 months
* Main organs function is normal
* Women of childbearing potential should agree to use and utilize an adequate method of contraception (such as intrauterine device，contraceptive and condom) throughout treatment and for at least 6 months after study is stopped；the result of serum or urine pregnancy test should be negative within 7 days prior to study enrollment，and the patients required to be non-lactating；Man participants should agree to use and utilize an adequate method of contraception throughout treatment and for at least 6 months after study is stopped
* Patients should participate in the study voluntarily and sign informed consent

Exclusion Criteria:

* 14 Days or more from the last cytotoxic therapy
* Patients participated in other anticancer drug clinical trials within 4 weeks or Patients participating in other clinical trials now
* Blood pressure unable to be controlled ideally by one drug(systolic pressure≥140 mmHg，diastolic pressure≥90 mmHg); Patients with Grade 1 or higher myocardial ischemia, myocardial infarction or malignant arrhythmias(including QTc≥470ms) and patients with Grade 3 or higher congestive heart failure (NYHA Classification)
* Patients with non-healing wounds or fractures
* Patients with drug abuse history and unable to get rid of or Patients with mental disorders
* History of immunodeficiency
* Patients with concomitant diseases which could seriously endanger their own safety or could affect completion of the study according to investigators' judgment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2017-09-13 (Actual); Primary Completion 2021-05-23 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
The maximum tolerated dose (MTD) of TQ-B3395 | 48 weeks
  The highest dose at which no more than 33% of the subjects experience a dose-limiting toxicity (DLT) during treatment
The type of dose-limiting toxicity(ies) (DLT[s]) of TQ-B3395 | For 4 weeks for DLTs.
  Subjects within 28 days after treatment appear the following toxicity reaction relate to the drug ：II °or above of kidney damage，III °or above of non-hematological toxicity,IV°hematological toxicity ,Neutropenia associated with fever
Pharmacokinetics of TQ-B3395 (in whole blood):Peak Plasma Concentration(Cmax) | up to 28 Days (endpoint when the two consecutive time points of blood drug concentration <150 DPM/mL)
  Peak Plasma Concentration(Cmax),Cmax in ng/mL.In the study of single-dose, full PK profiles will be obtained at H0/H1/H2/H3/H4/H8/H11/H24/H34/H48/H58/H72（H means Hour）.In the study of multiple-dose,full PK profiles will be obtained at D0/D1/D4/D7/D10/D14/D21（D means Day）.
Pharmacokinetics of TQ-B3395 (in whole blood):Peak time（Tmax） | up to 28 Days (endpoint when the two consecutive time points of blood drug concentration <150 DPM/mL)
  Peak time（Tmax）,Tmax in h.In the study of single-dose, full PK profiles will be obtained at H0/H1/H2/H3/H4/H8/H11/H24/H34/H48/H58/H72（H means Hour）.In the study of multiple-dose,full PK profiles will be obtained at D0/D1/D4/D7/D10/D14/D21（D means Day）
Pharmacokinetics of TQ-B3395 (in whole blood):Half life（t1/2） | up to 28 Days (endpoint when the two consecutive time points of blood drug concentration <150 DPM/mL)
  Half life（t1/2）,t1/2 in h.In the study of single-dose, full PK profiles will be obtained at H0/H1/H2/H3/H4/H8/H11/H24/H34/H48/H58/H72（H means Hour）.In the study of multiple-dose,full PK profiles will be obtained at D0/D1/D4/D7/D10/D14/D21（D means Day）
Pharmacokinetics of TQ-B3395 (in whole blood):Area under the plasma concentration versus time curve (AUC) | up to 28 Days (endpoint when the two consecutive time points of blood drug concentration <150 DPM/mL)
  Area under the plasma concentration versus time curve (AUC), AUC in ng.h/mL.In the study of single-dose, full PK profiles will be obtained at H0/H1/H2/H3/H4/H8/H11/H24/H34/H48/H58/H72（H means Hour）.In the study of multiple-dose,full PK profiles will be obtained at D0/D1/D4/D7/D10/D14/D21（D means Day）
Pharmacokinetics of TQ-B3395 (in whole blood):Clearance（CL） | up to 28 Days (endpoint when the two consecutive time points of blood drug concentration <150 DPM/mL)
  Clearance（CL）,CL in L/h.In the study of single-dose, full PK profiles will be obtained at H0/H1/H2/H3/H4/H8/H11/H24/H34/H48/H58/H72（H means Hour）.In the study of multiple-dose,full PK profiles will be obtained at D0/D1/D4/D7/D10/D14/D21（D means Day）

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | each 56 days up to intolerance the toxicity or PD (up to 24 months)

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided